CLINICAL TRIAL: NCT02829450
Title: Home-based Ultrafiltration for Congestive Heart Failure: Impact on Survival, Hospitalizations Rate, Quality of Life, Peritoneal Membrane Characteristics and Residual Renal Function With Different Treatment Modes
Brief Title: Peritoneal Ultrafiltration to Treat Congestive Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SOR-110-15-CTIL
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Kidney Disease; Congestive Heart Failure
Keywords: peritoneal ultrafiltration; congestive heart failure; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PD: Patients with CHF and chronic renal disease which started the treatment with peritoneal ultrafiltration.
  The patients will be follow up every 3 months for assesment of symptoms, QOL questionary, routine blood and urine tests and also for assesment of residual renal function and peritoneal membrane function: monitoring of clinical symptoms of fluid overload, hospital admissions, UF rate, peritoneal membrane damage parameters (cell-free DNA in peritoneal effluent, peritoneal equilibration test) and residual renal function markers (eGFR creatinine or cystatin C based , KT/V, urinary markers) at the start of the treatment, each 3 months during the treatment and at each change of prescription. Complications of all kinds will be recorded.
  Interventions: Other: peritoneal ultrafiltration
- Control: Patients with CHF and chronic renal disease which preferred to continue their regular treatment or choose other then peritoneal ultrafiltration type of renal replacement therapy (data from medical records): clinical symptoms of fluid overload, hospital admissions, urine volume,residual renal function markers (eGFR creatinine)

INTERVENTIONS:
Other: peritoneal ultrafiltration — Peritoneal fluids should be inserted intraperitoneally for several hours dwell
  Groups: PD

SUMMARY:
The purpose of this study is to determine whether the treatment of peritoneal ultrafiltration can improve survival and quality of life of refractory congestive heart failure with special accent on preserving residual renal function and peritoneal membrane characteristics/

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is the leading cause of acute hospital admissions. The morbidity associated with this condition presents a major health and economic challenge, which is anticipated to increase in the aging of population especially in developed countries.

Peritoneal dialysis (PD) in patients with diuretic resistant cardio-renal syndrome type 2 enables low-molecular weight solute clearance and ultrafiltration (UF) without serious hemodynamic changes, which makes this modality attractive for chronic CHF treatment . The key practical advantage of PD is that the patient can be treated at home, with treatment adjustment in accordance with his current condition. The additional advantages are: continuous UF, flexible schedule, no need for devices or anticoagulation, no need for medical staff.

Despite the fact that there was no significant improvement of survival in CHF patients treated by PD, as compared to regular treatment, improvement of symptoms, physical performance, quality of life , biochemical profile, and significant decrease in hospitalization rate have been reported.

PD has a number of both theoretical and practical advantages for extending treatment in CHF patients, but there is little experience in this field and limited knowledge regarding its influence on peritoneal membrane and renal function in patients with moderate renal failure.

Aims of the study:

1. primary aim - to find out if there is survival benefit on PD treatment, reduced hospitalization rate and improved QOL, to compare the functional outcomes of CHF patients 1 year before dialysis treatment and on PD treatment with different types of PD fluids
2. secondary aim - to choose the optimal type of dialysis treatment in term of effective UF, preservation of peritoneal membrane and residual renal function.

Research question: Whether UF improves survival and QOL in patients with severe CHF. What are the modes of PD and HD treatment ensuring the least possible negative impact on peritoneal membrane and residual renal function? Research hypothesis: UF improves survival and QOL in patients with severe CHF. Low glucose dialysis solutions are preferable treatment for CHF patient on PD for preservation of residual renal function and peritoneal membrane characteristics.

Possible risks preventing: early peritoneal membrane failure and deterioration of renal function, symptoms of fluid overload and need for inpatient treatment.

Type of study: observational prospective Population: CHF patients referred to nephrologist for home-based UF (PD) or medical or hemodialysis treatment

Inclusion criteria:

* diagnosis of heart failure NYHA 3-4 on maximal treatment with evidence of diuretic resistance and repeated hospital admissions due to fluid overload (at least 2 in previous 3 months)
* evidence of CKD stage 3-4
* agreement to place dialysis catheter in the peritoneal cavity for PD treatment or IV access for hemodialysis
* available medical records 1 year before dialysis treatment

Exclusion criteria:

* unstable hemodynamic or respiratory condition
* need for vasopressor support
* patient refusal
* lack of family support or housing conditions needed for PD treatment
* evidence of active kidney disease (obstructive uropathy, glomerulonephritis, vasculitis etc.) at recruitment to the study Accrual rate: 10 -20 patients per year, 40-80 patient overall Enrolment mode: The patients will be referred to peritoneal dialysis center by treating nephrologist or cardiologist. After identification and approval of candidate by dialysis nurse, the incident patients who meet the inclusion criteria, will be referred for peritoneal catheter insertion.

Intervention: PD catheter insertion by nephrologist or surgeon and PD treatment by dialysis fluids in according to clinical needs of the patient. Monitoring of clinical symptoms of fluid overload, hospital admissions, UF rate, peritoneal membrane damage parameters (cell-free DNA in peritoneal effluent, peritoneal equilibration test) and residual renal function markers (eGFR creatinine based , KT/V, urinary markers , PET) at the start of the treatment, each 3 months during the treatment and at each change of prescription. Complications of all kinds will be recorded.

Comparison group: CHF patients referred to nephrologist for home-based UF (PD) treatment and who preferred to continue conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of heart failure NYHA 3-4 on maximal treatment with evidence of diuretic resistance and repeated hospital admissions due to fluid overload (at least 2 in previous 3 months)
* evidence of CKD stage 3-4
* agreement to place dialysis catheter in the peritoneal cavity for PD treatment or IV access for hemodialysis
* available medical records 1 year before dialysis treatment

Exclusion Criteria:

* unstable hemodynamic or respiratory condition
* need for vasopressor support
* patient refusal
* lack of family support or housing conditions needed for PD treatment
* evidence of active kidney disease (obstructive uropathy, glomerulonephritis, vasculitis etc.) at recruitment to the study
* contraindications for peritoneal ultrafiltration treatment (active intraabdominal or abdominal wall inflammatory process, morbid obesity, multiple abdominal surgery in the past)
* non compliance with treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with chronic kidney disease and congestive heart failure refractory to medical therapy will be referred to peritoneal dialysis center by treating nephrologist or cardiologist. After identification and approval of candidate by dialysis nurse, the incident patients who meet the inclusion criteria, will be referred for peritoneal catheter insertion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 1 year

SECONDARY OUTCOMES:
ultrafiltration changes required change in peritoneal fluid prescription | 1 year
decrease in urine volume | 1 year
hospitalization for uncompensated heart failure | 1 year
complications, necessitating peritoneal catheter or hemodialysis catheter | 1 year
deterioration of renal function (every increasing in CKD stage) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marina Vorobiov, MD PhD, Principal Investigator — Soroka UMC
Locations (1):
- SorokaUMC, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meguid El Nahas A, Bello AK. Chronic kidney disease: the global challenge. Lancet. 2005 Jan 22-28;365(9456):331-40. doi: 10.1016/S0140-6736(05)17789-7. PMID 15664230
- [Background] Davies S, Lally F, Satchithananda D, Kadam U, Roffe C. Extending the role of peritoneal dialysis: can we win hearts and minds? Nephrol Dial Transplant. 2014 Sep;29(9):1648-54. doi: 10.1093/ndt/gfu001. Epub 2014 Feb 10. PMID 24520118
- [Background] Cnossen TT, Kooman JP, Krepel HP, Konings CJ, Uszko-Lencer NH, Leunissen KM, van der Sande FM. Prospective study on clinical effects of renal replacement therapy in treatment-resistant congestive heart failure. Nephrol Dial Transplant. 2012 Jul;27(7):2794-9. doi: 10.1093/ndt/gfr756. Epub 2012 Apr 6. PMID 22492829
- [Background] Hall MJ, Levant S, DeFrances CJ. Hospitalization for congestive heart failure: United States, 2000-2010. NCHS Data Brief. 2012 Oct;(108):1-8. PMID 23102190
- [Background] Wankowicz Z, Prochnicka A, Olszowska A, Baczynski D, Krzesinski P, Dziuk M. Extracorporeal versus peritoneal ultrafiltration in diuretic-resistant congestive heart failure--a review. Med Sci Monit. 2011 Dec;17(12):RA271-81. doi: 10.12659/msm.882118. PMID 22129914
- [Background] Prochnicka A, Krzesinski P, Halas K, Dziuk M, Niemczyk S, Wankowicz Z. Diuretic-resistant congestive heart failure treated successfully with peritoneal ultrafiltration. Kardiol Pol. 2013;71(4):393-5. doi: 10.5603/KP.2013.0067. PMID 23788345
- [Background] Ishimoto Y, Mise N, Tanaka M, Sugahara M, Kanemitsu T, Kobayashi M, Uchida L, Kotera N, Tanaka S, Sugimoto T. Peritoneal dialysis combined with extracorporeal ultrafiltration in refractory heart failure: a case report. Perit Dial Int. 2013 Sep-Oct;33(5):582-3. doi: 10.3747/pdi.2012.00212. No abstract available. PMID 24133088
- [Background] Ramachandran K, Speer CG, Fiddy S, Reis IM, Singal R. Free circulating DNA as a biomarker of prostate cancer: comparison of quantitation methods. Anticancer Res. 2013 Oct;33(10):4521-9. PMID 24123025